CLINICAL TRIAL: NCT07165275
Title: Factors Associated With Health-related Quality of Life in Patients With Breast Cancer-Related Lymphedema Undergoing Prospective Surveillance
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Other Study IDs: SMC 2024-05-116-001; RS-2023-CC139237 (Other Grant/Funding Number: Ministry of Health & Welfare)
Record Dates: First submitted 2025-07-28; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Related Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer-related lymphedema (BCRL) is a chronic condition that affects more than 1 in 5 breast cancer survivors. It causes swelling, pain, and reduced arm function, which can significantly impact quality of life. This study aims to evaluate how breast cancer survivors perceive their swelling, and whether this perception aligns with actual physical measurements. The investigation will examine how this perception gap relates to quality of life. The findings may help inform the development of more personalized care strategies to support both the physical and emotional well-being of women living with BCRL.

DETAILED DESCRIPTION:
This study focuses on identifying factors that influence health-related quality of life (HRQoL) in women with breast cancer-related lymphedema (BCRL). Prior studies have shown that the subjective burden of swelling and psychological responses may affect HRQoL more than objective clinical severity. However, the role of perception-objective congruence-whether participants' awareness of swelling matches actual physical measurements-has not been well explored. The investigators will analyze the impact of this perception gap on functional and emotional outcomes. Participants will be grouped based on whether their perception of swelling aligns with objective limb volume measurements. HRQoL differences across these subgroups will be assessed using validated instruments. The goal is to provide evidence that will inform strategies to promote accurate symptom awareness, effective self-management, and better quality of life in BCRL survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral upper limb lymphedema related to breast cancer
* Patients who have completed the Lymphedema Quality of Life Questionnaire (LYMQOL)

Exclusion Criteria:

* malignant lymphedema
* history of palliative chemotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with unilateral upper limb lymphedema related to breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Lymphedema Quality of Life Questionnaire (LYMQOL-Arm) | baseline
  Health Related Quality of Life(HRQoL) was assessed using the Lymphedema Quality of Life Questionnaire(LYMQOL), which comprises four domains: function (three items), appearance (five items), symptoms (six items), and mood (six items), scored on a 4-point Likert scale (1-4; higher scores indicate greater impairment). The domain scores were calculated as the average of the scores for all items within each domain. The LYMQOL also includes a single overall QoL item, which is scored on a scale from 0 (poor) to 10 (excellent)

SECONDARY OUTCOMES:
1. Age | baseline
  Demographic data
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
2. Sex | baseline
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
3. Body Mass Index (BMI) | baseline
  Demographic data Weight and height will be combined to report BMI (kg/m2)
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
4. Place of residence | baseline
  Demographic data
  (1) Metropolitan area, (2) Non- metropolitan area
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
5. Careers | baseline
  Demographic data Careers: Yes/No
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
6. Marital status | baseline
  Demographic data (0) Unmarried (Single/Widowed/Divorced), (1) Married
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
7. Number of comorbidities | baseline
  Demographic data
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
1. Time since breast cancer surgery | baseline
  data regarding cancer surgery and treatment
  1. Time since breast cancer surgery : years
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
2. Breact cancer stage | baseline
  data regarding cancer surgery and treatment Breact cancer stage : AJCC stage
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
3. Chemotherapy | baseline
  data regarding cancer surgery and treatment 3. Chemotherapy : Yes/No
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
4. Radiotherapy | baseline
  data regarding cancer surgery and treatment 4. Radiotherapy : Yes/No
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
5. Hormone therapy | baseline
  data regarding cancer surgery and treatment 5. Hormone therapy : Yes/No
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
1. Time since lymphedema diagnosis | baseline
  Lymphedema factors (medical records)
  1. Time since lymphedema diagnosis : years
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
2. Lymphedema in dominant hand | baseline
  Lymphedema factors (medical records) 2. Lymphedema in dominant hand : Yes/No
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
3. Lymphedema location | baseline
  Lymphedema factors (medical records) 3. Lymphedema location : Localized/Whole-arm
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
4. Complex Decongestive therapy | baseline
  Lymphedema factors (medical records) 4. Complex Decongestive therapy : Yes/No
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
5. perometer | baseline
  Lymphedema factors (medical records) 5. Limb volume was measured by perometer (Perometer®, Pero-System, Germany) : A perometer is a medical device used to measure limb volume accurately and non-invasively. It employs infrared light beams or optoelectronic sensors to scan the circumference of an extremity, such as an arm or leg, and calculates the overall volume based on these measurements. This tool is commonly used to assess swelling in conditions like lymphedema and to monitor changes over time.
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
1. Physical activity level | baseline
  Lymphedema factors (patient-reported)
  1. Physical activity level : Patient self-reported physical activity level categorized as limited in activities of daily living, not limited in activities of daily living, or able to participate in sports.
  Data collected through questions asked during clinical visits. All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
2. Lymphedema factors (patient-reported) | baseline
  Lymphedema factors (patient-reported) 2. Self-care adherence : Patient self-reported adherence to wearing compression stockings categorized as not wearing, wearing occasionally, or wearing regularly (including non-prescribed use).
  Data collected through questions asked during clinical visits. All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.
3. Subjective swelling severity | baseline
  Lymphedema factors (patient-reported) 3. Subjective swelling severity : Patient-rated swelling severity of the right/left arm on a numeric rating scale from 0 to 10, where 0 indicates no swelling and 10 indicates extremely severe swelling. Higher scores indicate worse
  Data collected via a survey asking, "How much do you think your right/left arm is swollen?".
  All anonymized clinical data were extracted from medical records in the Clinical Data Warehouse.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Republic of Korea, South Korea